CLINICAL TRIAL: NCT01441479
Title: Strep A Fluorescent Immunoassay and Analyzer Field Study
Status: Completed | Type: Observational
Sponsor: Quidel Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-0142-01
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2012-12

CONDITIONS: Strep Throat
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: In Vitro Diagnostic Device aid in diagnosing

SUMMARY:
The purpose of this study is to demonstrate the ability of the Strep A Fluorescent Immunoassay Analyzer to accurately detect a throat swab specimen for the presence or absence of Strep A when compared to culture.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects three (3) years of age or older

Must currently be exhibiting one or more of the following symptoms characteristic of pharyngitis

* Extreme sore throat
* Redness of the posterior pharyngeal wall
* Difficulty Swallowing
* Fever, >38.7C (100F) at presentation or within past 24 hours
* Pharyngeal exudate
* Tender cervical lymphadenopathy
* Absence of cough or other upper respiratory symptoms

Exclusion Criteria:

* Subjects currently under treatment with antibiotics are not to be included in this study.
* At clinical sites requiring informed consent, unable to understand and consent to participation; for minors this includes parent or legal guardian.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects must be greater than 3 years of age and exhibiting symptoms characteristic of pharyngitis, possibly Group A Streptococcus.
Sampling Method: Non-Probability Sample
Enrollment: 1282 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Streptococcus Group B identification | Immediate
  The purpose of this study was to identify via immunofluorescence technology, Group A Streptococcus, which was successfully done.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Best Medical Group, Phoenix, Arizona
  - La Costa Pediatrics, Carlsbad, California
  - La Jolla Pediatrics, San Diego, California
  - Teena Hughes, Tampa, Florida
  - FastER Urgent Care, Morris Plains, New Jersey
  - Twelve Corners Pediatrics, Rochester, New York
  - Advanced Pediatrics, Vienna, Virginia